CLINICAL TRIAL: NCT05287971
Title: Improving Standard of Care Lifestyle Support for Stage III NSCLC Cancer Patients
Brief Title: Standard of Care Lifestyle Support for Stage III NSCLC Patients
Acronym: PERCUSSION
Status: Withdrawn | Type: Observational
Why Stopped: Never started
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PERCUSSION
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle advice — Patients will receive lifestyle advice regarding nutricion and exercise and will be monitored with regard to exercise and vital signs.

SUMMARY:
Offering an early-initiated supportive care program to stage III NSCLC patients to prevent deterioration of performance status and increase compliance of patients that complete chemoradiation as well as the patients receiving 12 months of durvalumab.

DETAILED DESCRIPTION:
In inoperable Stage III Non-Small Cell Lung Cancer (NSCLC), consolidation immune checkpoint inhibition with the PD-L1 inhibitor durvalumab, given within 6 weeks after completion of concurrent platinum-based chemoradiotherapy (CCRT) for 12 months results in remarkable improvement of 3-year overall survival rates (57% vs 43.5%). This tri-modal therapy has become the new standard of care. Unfortunately, the tri-modal therapy frequently causes adverse events such as fatigue and, to a much lesser degree, cough, dyspnea and pneumonitis, resulting in treatment cessation in 15% - 53% of the patients (15%) (53%). For the most optimal overall survival (OS) and disease-free survival (DFS), compliance to the full treatment regimen, i.e. in the ideal situation 100% of patients completing their full course of CCRT and receiving durvalumab for one year, is expected to have significant and relevant beneficial effects. Optimizing patients' fitness is essential in order to handle the tough full treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of adequately staged (according to standard practice using chest-CT, FDG-PET, brain imaging MRI/CT) NSCLC
* Participant is willing and able to give informed consent for participation in the trial
* Aged 18 years or above
* Scheduled to receive one of the following two therapeutic strategies:

  * Concurrent chemotherapy and radiotherapy with photons (60 Gy in 30 fractions of 2 Gy) followed by durvalumab in patients with stage III NSCLC
  * Concurrent chemotherapy and radiotherapy with protons (60 Gy in 30 fractions of 2 Gy) followed by durvalumab in patients with stage III NSCLC
* Able and willing to comply with all trial requirements

Exclusion Criteria:

* Mixed non-small cell lung cancer with other histology such as small cell lung cancer
* Not able to comply with the study protocol
* Less than 18 years old
* Pregnancy or not able to comply with adequate contraception in women with child baring potential
* Previous radiotherapy to the chest for benign or malignant conditions, including radiation for breast cancer
* Previous malignancy treated with chemotherapy, immune therapy or radiotherapy (irrespective of when this happened)
* Previous malignancies treated with surgery only are allowed if 2 years or more before inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III NSCLC who are eligible for curative intent concurrent chemotherapy and radiotherapy as well as willing to adhere to the study protocol will be enrolled in the study. They receive standard radiotherapy (60 Gy in 30 fractions of 2 Gy) with photons (group 1) or protons (group 2) according to the standard of care. Eligible patients will thereafter receive standard durvalumab immune therapy for 12 months. Eligibility criteria for this study are therefore similar to those for standard of care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Compliance | 12 months
  Compliance to CCRT and durvalumab treatment

SECONDARY OUTCOMES:
Percentage adhering advice | 12 months
  Improving standard of care lifestyle support by measuring % patients successfully adhering to the dietary, exercise, smoking advice
Perctenage use of watch | 12 months
  Improving standard of care lifestyle support by measuring % use of the watch (and app)
Percentage dysphagia | 12 months
  Improving standard of care lifestyle support by measuring % grade 3 dysphagia and odynophagia
Percentage dyspnea | 12 months
  Improving standard of care lifestyle support by measuring % grade 2 dyspnea
Percentage hospitalization | 12 months
  Improving standard of care lifestyle support by measuring % hospitalization for (treatment-related) complications + specification (from start until 6 weeks after radiotherapy)
Standard of care lifestyle support | 12 months
  Measuring match between lifestyle advice and personal circumstances by questionnaire
Barriers | 12 months
  Measuring adherence of barriers and facilitators in lifestyle support by questionnaire
Proton/photon | 12 months
  Improving standard of care lifestyle support by measuring the difference between proton and photon therapy i the above mentioned outcome
Durvalumab | 12 months
  Improving standard of care lifestyle support by measuring % patients receiving durvalumab
Quality of life questionnaire | 12 months
  Improving standard of care lifestyle support by measuring the quality of life by EORTC QLQ-C30/-LC13

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro; Karen Zegers, MD, PhD, Principal Investigator — Maastro; Lizza Hendriks, MD, PhD, Principal Investigator — Maastricht University Hospital (MUMC+); Cheryl Roumen, PhD, Study Director — Maastro

IPD SHARING:
Plan to Share IPD: No